CLINICAL TRIAL: NCT06363461
Title: A Randomized, Vehicle-Controlled, Parallel Group Study of Topical TDM-180935 to Evaluate the Preliminary Efficacy, Safety, Tolerability, and Pharmacokinetics in Atopic Dermatitis Patients
Brief Title: Study of TDM-180935 in Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technoderma Medicines Inc. (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 239-13851-202
Record Dates: First submitted 2024-04-03; First posted 2024-04-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TDM-180935 topical ointment 1.0% (Experimental): Daily dose of 1.0% of TDM-180935 topical ointment
  Interventions: Drug: TDM-180935 topical ointment 1.0%
- TDM-180935 topical ointment 2.0% (Experimental): Daily dose of 2.0% of TDM-180935 topical ointment
  Interventions: Drug: TDM-180935 topical ointment 2.0%
- TDM-180935 topical vehicle ointment 1 (Placebo Comparator): Daily dose of placebo color matched to TDM-180935 topical ointment 1.0%
  Interventions: Drug: TDM-180935 topical vehicle ointment 1
- TDM-180935 topical vehicle ointment 2 (Placebo Comparator): Daily dose of placebo color matched to TDM-180935 topical ointment 2.0%
  Interventions: Drug: TDM-180935 topical vehicle ointment 2

INTERVENTIONS:
Drug: TDM-180935 topical ointment 1.0% — TDM-180935 topical ointment 1.0%
  Arms: TDM-180935 topical ointment 1.0%
Drug: TDM-180935 topical ointment 2.0% — TDM-180935 topical ointment 2.0%
  Arms: TDM-180935 topical ointment 2.0%
Drug: TDM-180935 topical vehicle ointment 1 — TDM-180935 topical vehicle ointment 1
  Arms: TDM-180935 topical vehicle ointment 1
Drug: TDM-180935 topical vehicle ointment 2 — TDM-180935 topical vehicle ointment 2
  Arms: TDM-180935 topical vehicle ointment 2

SUMMARY:
Randomized, Vehicle-controlled, Parallel Group Study of TDM-180935 in Atopic Dermatitis Patients

DETAILED DESCRIPTION:
Protocol 239-13851-202 is a Phase 2a study entitled "A Randomized, Vehicle-Controlled, Parallel Group Study of Topical TDM-180935 to Evaluate the Preliminary Efficacy, Safety, Tolerability, and Pharmacokinetics in Atopic Dermatitis Patients". Eligible subjects (24) in the randomized portion of the study will be randomized (2:2:1:1) to 1 of the 4 groups (low dose vs high dose vs placebo 1 vs placebo 2) and treated for 8 weeks. Eligible subjects (6) in the PK (pharmacokinetics) cohort will be treated with the high dose in an open label fashion.

ELIGIBILITY:
Inclusion Criteria:

1. A) Patient is a male ≥ 18 years old at Visit 1/Screening. B) Patient is a post-menopausal or surgically sterile female ≥ 18 years old at Visit 1/Screening.
2. Patient has provided written informed consent.
3. Male patients who are sexually active with a female partner and are not surgically sterile must use a highly effective method of birth control as described in the informed consent form. Note: Male patients must refrain from sperm donation for at least 90 days after application of their last dose of IP (investigational product).
4. Patient has active mild or moderate AD with a modified-Eczema Area and Severity Index (m-EASI) score of 5-16 and a history of AD duration ≥ 2 years.
5. Patient has an AD body surface area (BSA) between 3 and 12% in the area to be treated (excluding head/neck, hands/feet, genitalia, and intertriginous areas) at Baseline.
6. Patient is willing and able to apply the IP(s) as directed, comply with study instructions (including avoiding direct sunlight exposure to the areas of IP application), and commit to all follow-up visits for the duration of the study. Note: The use of topical sunscreen is permitted provided the patient has used the sunscreen previously and it does not contain any prohibited medications/ingredients.
7. Patient, in the investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation or exposes the patient to an unacceptable risk by study participation.
8. Patient agrees to apply a bland moisturizer as directed for the duration of the study.
9. Patient has normal renal and hepatic function as determined by the Visit 1/Screening laboratory results in the opinion of the investigator.
10. [For PK Cohort Only] Patient is a non-smoker, defined as not having smoked or used any form of tobacco or non-tobacco products containing nicotine in more than 6 months before Visit 2/Baseline.
11. [For PK Cohort Only] Patient has a body mass index (BMI) of 19 to 32 kg/m2 inclusive and body weight not less than 50 kg at Visit 1/Screening.

Exclusion Criteria:

1. Patient has any dermatological disorders of the skin within 20 cm of the areas to be treated with the possibility of interfering with the application of the IP or examination method, such as fungal or bacterial infections, psoriasis, folliculitis, notable scarring (linear scar > 2.5 cm, etc.), or skin atrophy at Visit 2/Baseline.
2. Patient has any skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the IP or requires use of interfering topical, systemic, or surgical therapy at Visit 2/Baseline.
3. Patient has any visible inflammatory skin disease, injury, or condition of their skin that could compromise patient safety and/or interfere with the evaluation of local or systemic assessments performed during the study.
4. Patient has a known or suspected malignancy at Visit 2/Baseline excluding basal cell skin cancer unless it is associated with the area to be treated per Exclusion Criterion no. 1.
5. Patient has a positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
6. Patient has any condition, which, in the investigator's opinion, would make it unsafe for the patient to participate in this study, including clinically significant abnormal laboratory, or 12-lead electrocardiogram (ECG) findings during the screening period or Visit 2/Baseline prior to dosing of the IP.
7. Patient has a hospital admission or major surgery within 30 days prior to Visit 2/ Baseline or planned for during the study.
8. Patient is currently enrolled in an investigational drug, biologic, or device study.
9. Patient has used an investigational drug, investigational biologic, or investigational device treatment within 30 days or 5 half-lives, whichever is longer, prior to Visit 2/Baseline.
10. Patient has a history of prescription drug abuse, or illicit drug use within 6 months prior to Visit 1/Screening.
11. Patient has a history of alcohol abuse according to medical history within 6 months prior to Visit 1/Screening.
12. Patient has a positive screen for alcohol or drugs of abuse at Visit 1/Screening or Visit 2/Baseline. Note: Patients with a positive drug screen believed by the investigator to be the result of medically appropriate prescription medication use can be enrolled with Medical Monitor approval.
13. Patient has used topical cosmetic (excluding bland moisturizers), herbal, over-the- counter (OTC) or prescription products within areas to be treated within 2 weeks prior to dosing at Visit 2/Baseline.
14. Patient has used systemic prescription treatment for AD or that in the opinion of the investigator may affect the patient's AD (examples include, but are not limited to PDE4 (Phosphodiesterase-4) inhibitors, corticosteroids, immunomodulators, antimetabolites, antibiotics, retinoids, etc.) within 4 weeks prior to Visit 2/Baseline. Note: systemic corticosteroids do not include intranasal, inhaled, or ophthalmic corticosteroids for the management of allergies, pulmonary disorders, or other conditions.
15. Patient has used systemic biologic therapy (i.e., dupilumab) for AD or that in the opinion of the investigator may affect the patient's AD within 5 half-lives of the biologic therapy prior to Visit 2/Baseline.
16. Patient has been diagnosed with COVID-19 (Coronavirus Disease of 2019) within 4 weeks of Visit 1/Screening.
17. Patient is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
18. Patient has previously been treated with the IP.
19. Patient has a history of sensitivity to any of the ingredients in the IP.
20. Patient has ongoing or recent history of any other uncontrolled and/or clinically significant systemic disease or condition which, in the investigator's opinion, should exclude participation in the study.
21. [For PK Cohort Only] Patient has a donation or blood collection of more than 1 unit (approximately 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to Visit 2/Baseline.
22. [For PK Cohort Only] Patient has used systemic prescription medications, herbal (including St John's Wort, herbal teas and garlic extracts) supplements within 14 days prior to dosing at Visit 2/Baseline.
23. [For PK Cohort Only] Patient has used systemic OTC medications or vitamins within 7 days prior to dosing at Visit 2/Baseline. (Note: Use of acetaminophen at < 3g/day is permitted).
24. [For PK Cohort Only] Patient received a live or live attenuated vaccine within 4 weeks of dosing at Visit 2/Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 1. Patient is a male ≥ 18 years old
  2. Patient is a post-menopausal or surgically sterile female ≥ 18 years old
Enrollment: 24 (Actual)
Dates: Start 2024-04-13 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Change in m-EASI (modified Eczema Area and Severity Index) score | 8 weeks
  Collection of EASI (Eczema Area and Severity Index) results at week 8. The total m-EASI score may range from zero (0) to a maximum of 64.8, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Proportion of patients with a ≥ 2 point improvement in vIGA-AD score (validated Investigator's Global Assessment for Atopic Dermatitis score) | 8 weeks
  Collection of vIGA-AD score (validated Investigator's Global Assessment for Atopic Dermatitis score) at week 8. The vIGA-AD is a static morphological 5-point ordinal scale from 0 (clear) to 4 (severe).
Change in m-EASI (modified Eczema Area and Severity Index) score | 6 weeks
  Collection of EASI (Eczema Area and Severity Index) results at weeks 2, 4, and 6. The total m-EASI score may range from zero (0) to a maximum of 64.8, and higher scores mean a worse outcome.
Proportion of patients with a 50% improvement in m-EASI (modified Eczema Area and Severity Index) score | 8 weeks
  Collection of EASI (Eczema Area and Severity Index) results at week 8. The total m-EASI score may range from zero (0) to a maximum of 64.8, and higher scores mean a worse outcome.
Proportion of patients with a 75% improvement in m-EASI (modified Eczema Area and Severity Index) score | 8 weeks
  Collection of EASI (Eczema Area and Severity Index) results at week 8. The total m-EASI score may range from zero (0) to a maximum of 64.8, and higher scores mean a worse outcome.
Proportion of patients with a 90% improvement in m-EASI (modified Eczema Area and Severity Index) score | 8 weeks
  Collection of EASI (Eczema Area and Severity Index) results at week 8. The total m-EASI score may range from zero (0) to a maximum of 64.8, and higher scores mean a worse outcome.
Change in BSA (body surface area) affected | 8 weeks
  Collection of BSA affected at weeks 2, 4, 6, and 8
Proportion of patients with a 4-point improvement from Baseline in WI-NRS (Worst Itch-Numeric Rating Scale) score | 8 weeks
  Collection of WI-NRS (Worst Itch-Numeric Rating Scale) score at week 8. The level of itching is described on an 11-point scale anchored at 0, representing "no itch" and 10, representing, "worst itch imaginable".

OTHER OUTCOMES:
Incidence (severity and causality) of any local and systemic AEs (adverse events) | 8 weeks
  Collection of adverse events
Number of patients with presence (and severity) of the following LSRs (local skin reactions): skin pigmentation (hyperpigmentation and hypopigmentation), edema, erosion,scaling, and burning/stinging | 8 weeks
  Collection of LSRs at weeks 2, 4, 6, and 8
Changes from Baseline in vital signs (temperature) | 8 weeks
  Collection of temperature at weeks 4 and 8
Changes from Baseline in vital signs (systolic and diastolic blood pressure) | 8 weeks
  Collection of systolic and diastolic blood pressure at weeks 4 and 8
Changes from Baseline in vital signs (heart rate) | 8 weeks
  Collection of heart rate at weeks 4 and 8
Changes from Baseline in vital signs (respiration rate) | 8 weeks
  Collection of respiration rate at weeks 4 and 8
Changes from baseline in clinical laboratory tests (including Blood Chemistries, Hematology, and Urinalysis) | 8 weeks
  Collection of safety lab results at weeks 4 and 8
Number of participants with abnormal ECG readings | 8 weeks
  Collection of ECGs at day1, week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Piacquadio, M.D., Study Director — Therapeutics Incorporated
Locations (7):
- United States (7):
  - Site 5, Rolling Meadows, Illinois
  - Site 8, Covington, Louisiana
  - Site 4, New Brighton, Minnesota
  - Site 7, Anderson, South Carolina
  - Site 3, Austin, Texas
  - Site 1, College Station, Texas
  - Site 2, Norfolk, Virginia